CLINICAL TRIAL: NCT05417594
Title: A Modular Phase I/IIa, Open-label, Multi-centre Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Ascending Doses of AZD9574 as Monotherapy and in Combination With Anti-cancer Agents in Patients With Advanced Solid Malignancies (CERTIS1)
Brief Title: Study of AZD9574 as Monotherapy and in Combination With Anti-cancer Agents in Participants With Advanced Solid Malignancies
Acronym: CERTIS1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8410C00001; 2023-504984-17-00 (Registry Identifier: CTIS (EU)); 2021-006227-17 (EudraCT Number)
Record Dates: First submitted 2022-05-20; First posted 2022-06-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Malignancies
Keywords: Poly ADP-ribose Polymerase inhibitor (PARPi); Anti-tumour; Breast cancer; Ovarian cancer; Fallopian tube cancer; Prostate cancer; Pancreatic cancer; Soft tissue disease; Glioma; Astrocytoma; Oliogodendroglioma; Solid tumours
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Glioma; Astrocytoma | interventions — Temozolomide; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Module 1 Part A: Dose escalation (Experimental): Participants with advanced/relapsed ovarian, breast, pancreatic, or prostate cancer who are deemed suitable for a PARPi will receive AZD9574 monotherapy at escalating cohorts.
  Interventions: Drug: AZD9574
- Module 1 Part B: Dose expansion (Experimental): Participants with breast cancer who are PARPi naive at doses determined in dose-escalation.
  Interventions: Drug: AZD9574
- Module 2 Part A: Dose escalation (Experimental): Participants with IDH 1/2-mutant glioma who are PARPi naive will receive AZD9574 and TMZ at escalating cohorts.
  Interventions: Drug: AZD9574; Drug: Temozolomide (TMZ)
- Module 3 Panel 1: AZD9574 monotherapy (Sweden only) (Experimental): Participants with advanced/relapsed HER2-negative breast, ovarian, prostate, or pancreatic cancer and expressing BRCA1m, BRCA2m, PALB2m, RAD51Cm or RAD51Dm.
  Interventions: Drug: AZD9574; Drug: [11C]AZ1419 3391
- Module 3 Panel 2: AZD9574 + TMZ (Sweden only) (Experimental): Participants with IDH 1/2-mutant glioma who are PARPi naive will receive AZD9574 and TMZ at escalating cohorts.
  Interventions: Drug: AZD9574; Drug: Temozolomide (TMZ); Drug: [11C]AZ1419 3391
- Module 3 Panel 3: AZD9574 monotherapy (Sweden only) (Experimental): Participants with breast cancer (without BM).
  Interventions: Drug: AZD9574; Drug: [11C]AZ1419 3391
- Module 4 Part A: Dose escalation (AZD9574 + T-DXd) (Experimental): Participants with advanced, unresectable, or metastatic solid tumours that are HER2-positive will receive a combination of AZD9574 and T-DXd at at escalating cohorts.
  Interventions: Drug: AZD9574; Drug: Trastuzumab Deruxtecan (T-DXd)
- Module 4 Part B : Dose expansion (AZD9574 + T-DXd) (Experimental): Participants with HER2-low/ultralow, HR positive breast cancer will receive a combination of different doses of AZD9574 and T-DXd at expanding cohorts.
  Interventions: Drug: AZD9574; Drug: Trastuzumab Deruxtecan (T-DXd)
- Module 5 Part A : Dose escalation (AZD9574 + Dato-DXd) (Experimental): Participants with advanced, unresectable, or metastatic solid tumours in different types of cancers will receive a combination of AZD9574 and Dato-DXd at escalating cohorts.
  Interventions: Drug: AZD9574; Drug: Datopotamab Deruxtecan (Dato-DXd)

INTERVENTIONS:
Drug: AZD9574 — Participants will receive AZD9574 orally.
Drug: Temozolomide (TMZ) — Participants will receive temozolomide orally.
  Arms: Module 2 Part A: Dose escalation; Module 3 Panel 2: AZD9574 + TMZ (Sweden only)
Drug: [11C]AZ1419 3391 — Participants will receive [11C]AZ1419 3391 intravenously.
  Arms: Module 3 Panel 1: AZD9574 monotherapy (Sweden only); Module 3 Panel 2: AZD9574 + TMZ (Sweden only); Module 3 Panel 3: AZD9574 monotherapy (Sweden only)
Drug: Trastuzumab Deruxtecan (T-DXd) — Participants will receive T-DXd intravenously.
  Arms: Module 4 Part A: Dose escalation (AZD9574 + T-DXd); Module 4 Part B : Dose expansion (AZD9574 + T-DXd)
Drug: Datopotamab Deruxtecan (Dato-DXd) — Participants will receive Dato-DXd intravenously.
  Arms: Module 5 Part A : Dose escalation (AZD9574 + Dato-DXd)

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of AZD9574 individually and in combination with anti-cancer agents in participants with advanced cancer that has recurred/progressed.

DETAILED DESCRIPTION:
This is a modular phase I/IIa, multi-centre, multi-part, open-label, dose escalation, and dose expansion study.

Approximately 695 participants will be enrolled and assigned to study treatments.

This study consists of individual modules each evaluating safety and tolerability.

* Core protocol which contains information applicable to all modules.
* Module 1 (AZD9574 monotherapy):

This module will include 235 participants:

* Part A (dose-escalation cohorts) will include participants with advanced/relapsed ovarian, breast, pancreatic or prostate cancer that are deemed suitable for a Poly ADP-Ribose Polymerase (PARPi) by the Investigator.
* Part B (dose-expansion cohorts):

This module will include up to 3 expansion cohorts with 30 participants in each:

* Cohort B1 will include participants with advanced/relapsed Human Epidermal Growth Factor Receptor 2 (HER2)-negative breast cancer participants with breast cancer gene (BRCA) mutated (BRCA1m, and BRCA2m), partner and localiser of the BRCA2 gene (PALB2) mutation (PALB2m), RAD51Cm or RAD51Dm, without evidence of untreated brain metastasis at baseline Magnetic Resonance Imaging (MRI) scan.
* Cohort B2 will include participants with advanced/relapsed HER2-negative breast cancer participants with BRCA1m, BRCA2m, PALB2m, RAD51Cm or RAD51Dm, who have either untreated or treated brain metastases that are not requiring immediate local therapy.

  * Up to of 20 participants may be required to get 12 evaluable participants in each cohort for food effect and Acid Reducing Agent (ARA) investigations.

    • Module 2 (AZD9574 in combination with temozolomide (TMZ): This module will include 75 participants for up to 12 cycles.
  * Part A (dose-escalation cohorts) will include participants with Isocitrate Dehydrogenase (IDH)-mutant glioma.

    • Module 3 (PET Sub-study: AZD9574 monotherapy [Panels 1 and 3], AZD9574 in combination with TMZ (Panel 2). This module will include 12 participants and is only applicable for Sweden.
  * Panel 1 (AZD9574 monotherapy) will include up to 8 participants with advanced/relapsed HER2-negative breast, ovarian, prostate, or pancreatic cancer and expressing BRCA1m, BRCA2m, PALB2m, RAD51Cm or RAD51Dm.
  * Panel 2 (AZD9574 + TMZ) will include up to 2 participants with IDH-mutant recurrent glioma.
  * Panel 3 (AZD9574 monotherapy) will include up to 2 participants with breast cancer (without BM).

    * Module 4 (AZD9574 in combination with Trastuzumab deruxtecan [T-DXd])

This module will include 265 participants (including backfills):

* Part A (dose escalation cohorts) will include participants with advanced, unresectable, or metastatic solid tumours that are HER2-positive.
* Part B (dose expansion cohorts) will include up to 4 cohorts with participants with HER2-low/ultralow, HR positive breast cancer. Approximately 30 response evaluable participants without brain metastases will be enrolled in each cohort and up to 10 additional participants with brain metastases (CNS cohort) may be enrolled in each cohort.

  * Module 5 (AZD9574 in combination with Datopotamab deruxtecan [Dato-DXd])

This module will include 105 participants (including backfills):

* Part A (dose escalation cohorts) will include participants with advanced, unresectable, or metastatic solid tumours in different types of cancers.
* Part B (dose expansion cohorts) may be added in the future amendment.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status (ECOG PS) with no deterioration over the previous 2 weeks.
* Progressive cancer at the time of enrollment.
* Adequate organ and marrow function.

Module 1:

Part A:

- Participants must have one of the following: (i) Histologically or cytologically confirmed relapsed advanced ovarian, fallopian tube or primary peritoneal cancer and evidence of a predicted loss of function germline or tumour mutation in one of the following homologous recombination repair genes: BRCA1, BRCA2, PALB2, RAD51C or RAD51D (ii) Histologically or cytologically confirmed HER2-negative carcinoma of the breast with recurrent locally advanced or metastatic disease and evidence of a predicted loss of function germline or tumour mutation in one of the following homologous recombination repair genes: BRCA1, BRCA2, PALB2, RAD51C, or RAD51D.

(iii) Histologically or cytologically confirmed advanced/metastatic castration-resistant prostate cancer (CRPC) and evidence of a predicted loss of function germline or tumour mutation in one of the following homologous recombination repair genes:BRCA1, BRCA2, PALB2, RAD51C, or RAD51D (d) Histologically or cytologically confirmed advanced/metastatic pancreatic cancer and evidence of a predicted loss of function germline or tumour mutation in one of the following homologous recombination repair genes: BRCA1, BRCA2, PALB2, RAD51C, or RAD51D.

* Must have evaluable disease.
* Must be suitable for treatment with a PARPi.
* Must be capable of eating a high fat meal and adhering to fasting restrictions.

Part B:

* Must have metastatic or recurrent locally advanced histologically or cytologically confirmed Human Epidermal growth factor Receptor 2 (HER2)-negative carcinoma of the breast and evidence of a predicted loss of function germline or tumour mutation.
* Must have at least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter.
* Participants who have received platinum chemotherapy for advanced breast cancer are eligible to enter the study provided there has been no evidence of disease progression during the platinum chemotherapy.
* Participants who have received prior platinum-based chemotherapy as neo-adjuvant/adjuvant treatment are eligible provided at least 12 months have elapsed between the last dose of platinum-based treatment and first dose of study intervention.

Module 2:

* Must be suitable for treatment with TMZ and have IDH1/2-mutant glioma.
* Should have progressive disease after prior radiation therapy and one prior line of alkylating chemotherapy for their disease.
* Recurrent disease must be evaluable by MRI.
* Female participants of childbearing potential (CBP) must have a negative pregnancy test result at screening and prior to each cycle administration of AZD9574 and TMZ.
* Adequate organ and marrow function.

Module 3:

Panel 1

* Must consent to provide mandated blood samples and archival/fresh tumour tissue for confirmatory tests of their cancer using central laboratory.
* Participants must have one of the following:

  1. Histologically or cytologically confirmed HER2-negative carcinoma of the breast with recurrent locally advanced or metastatic disease and evidence of a predicted loss of function germline or tumour mutation in BRCA1, BRCA2, PALB2, RAD51C, or RAD51D,
  2. Histologically or cytologically confirmed relapsed advanced ovarian, fallopian tube or primary peritoneal cancer and evidence of a predicted loss of function germline or tumour mutation in BRCA1, BRCA2, PALB2, RAD51C, or RAD51D
  3. Histologically or cytologically confirmed advanced/metastatic castration-resistant prostate cancer (CRPC) and evidence of a predicted loss of function germline or tumour mutation in in BRCA1, BRCA2, PALB2, RAD51C or RAD51D.
  4. Histologically or cytologically confirmed advanced/metastatic pancreatic cancer and evidence of a predicted loss of function germline or tumour mutation in in BRCA1, BRCA2, PALB2, RAD51C, or RAD51D.
* Participants must have evaluable disease: at least one measurable and/or non-measurable lesions per RECIST 1.1
* Must be refractory to standard therapy or for which no standard therapy exists.
* Any 2 participants in this panel must meet the following CNS criteria:

  1. Must have previously treated and progressing or untreated brain metastases confirmed by brain MRI at screening that do not need immediate local therapy.
  2. Should have stable neurological function for ≥ 14 days prior to signing the main study ICF.
  3. If receiving steroids, the dose should be stable or decreasing for ≥ 14 days prior to signing the main study ICF.

Panel 2

* Must be suitable for treatment with TMZ and have IDH1/2-mutant glioma.
* Should have progressive disease after prior radiation therapy and one prior line of alkylating chemotherapy for their disease.
* Recurrent disease must be evaluable by MRI and at least 1 tumour of > 1cm diameter detected on MRI.
* Formalin-fixed, paraffin-embedded (FFPE) tumour sample from the primary cancer must be available for central testing
* Adequate organ and marrow function (in the absence of transfusions or growth factor support within 14 days prior to enrolment)

Panel 3

* Must consent to provide mandated blood samples and archival/fresh tumour tissue for confirmatory tests of their cancer using central laboratory.
* Must have histologically or cytologically confirmed HER2-negative carcinoma of the breast with recurrent locally advanced or metastatic disease and evidence of a predicted loss of function germline or tumour mutation in in BRCA1, BRCA2, PALB2, RAD51C or RAD51D .
* Must have evaluable disease: at least one measurable and/or non-measurable lesions per RECIST 1.1 .
* Must be refractory to standard therapy or for which no standard therapy exists.

Module 4:

Part A:

* Must have the following HER2 status:

  1. Breast cancer must be IHC 3+ or IHC 2+/ISH-positive or IHC 2+/ISH-negative or IHC 1+ as determined by local testing using current American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) guidelines for scoring HER2 + breast cancer.
  2. Gastric cancer should be IHC 3+ or IHC 2+/ISH-positive based on local tissue testing results.
  3. Participants with non-breast and non-gastric cancers must have HER2-overexpression (IHC 3+ or IHC 2+; as determined by local testing using current ASCO-CAP guidelines for gastric IHC scoring).
  4. Participants with NSCLC will also be eligible based on the presence of a HER2activating mutation.
* Must have progressed following at least one prior systemic treatment and not more than 2 prior lines of cytotoxic therapy for metastatic or advanced disease and have no satisfactory alternative treatment option.
* Should have unresectable, or metastatic disease based on most recent imaging. The following tumour types are eligible for this study: Breast cancer, Non-Small Cell Lung Cancer, Colorectal Cancer, Bladder Cancer, Ovarian Cancer, Gastric Cancer, and Other tumour types ( unresectable or metastatic biliary tract cancer, cervical cancer, endometrial cancer, and pancreatic adenocarcinoma).
* Adequate organ and marrow function (in the absence of transfusions or growth factor support) within 14 days prior to the first dose of study intervention.
* Left ventricular ejection fraction (LVEF) ≥ 50% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before start of treatment.
* Must have at least one lesion not previously irradiated (or with evidence of disease progression following radiation).
* Non-sterilised male participants who are sexually active with a female partner of CBP must use a condom with spermicide from screening to approximately 6 months after the last dose of study intervention.
* Male participants must refrain from fathering a child or donating sperm during the study and for approximately 6 months after the last dose of study intervention.

Part B - All participants:

* Histologically documented unresectable or metastatic breast cancer.
* Metastatic or recurrent locally advanced unresectable histologically or cytologically confirmed HER2-low or HER2-ultralow breast carcinoma.
* No prior chemotherapy for locally advanced unresectable or metastatic breast cancer.

Part B - Participants with brain metastases:

* Stable neurological function for ≥ 14 days prior to signing the main study ICF.
* If receiving steroids, the dose should be stable or decreasing for ≥ 14 days prior to signing the main study ICF.
* Must not have progressing or untreated (stable or progressing) brain metastases.

Part B - Participants in CNS cohort:

- Untreated brain metastases, previously treated and stable or progressing brain metastases on screening contrast brain MRI/CT scan, not needing immediate local therapy.

Module 5 :

* Should have unresectable, or metastatic disease based on most recent imaging. The following tumour types are eligible for this study: TNBC, Endometrial cancer, Ovarian Cancer and CRPC.
* Must have progressed following at least one prior systemic treatment for metastatic or advanced disease and have no satisfactory alternative treatment option.
* Must have at least one lesion, not previously irradiated that can be accurately measured at baseline as ≥ 10 mm in the longest diameter.
* Non-sterilised male participants who are sexually active with a female partner of CBP must use a condom with spermicide from screening to approximately 4 months after the last dose of study.
* Male participants must refrain from fathering a child or donating sperm during the study and for approximately 4 months after the last dose of study intervention.
* Adequate organ and marrow function (in the absence of transfusions or growth factor support) within 14 days prior to the first dose of study intervention.

Modules 1, 2 and 3:

* Female participants of CBP:

  1. Must have a negative pregnancy test result at screening and prior to each cycle of study treatment.
  2. If sexually active with a non-sterilised male partner, must use at least one highly effective method of birth control plus a barrier method from screening to approximately 6 months after the last dose of study treatment.
* Female participants must not breastfeed and must not donate or retrieve ova for their own use from screening to approximately 6 months after the last dose of study treatment.
* Non-sterilised male participants who are sexually active with a female partner of CBP must use a condom with spermicide from screening to approximately 3 months after the last dose of study intervention.
* Female partners of male participants should use at least one highly effective method of contraception from screening to approximately 3 months after the last dose of study intervention of the male participant.
* Male participants must refrain from fathering a child or donating sperm from the start of study intervention and for approximately 3 months after the last dose of study intervention.

Modules 4 and 5:

* Female participants of CBP:

  1. Must have a negative pregnancy test result at screening and prior to each cycle of study intervention.
  2. If sexually active with a non-sterilised male partner, must use at least one highly effective method of birth control in combination with one effective method (male condom plus spermicide) from screening until approximately 7 months after the last dose of study intervention.
* Female participants must not breastfeed and must not donate or retrieve ova for any use from screening to approximately 7 months after the last dose of study intervention.
* Participants must provide an existing FFPE tumour sample for retrospective, tissue-based IHC testing in a central laboratory to determine HER2 expression and other correlatives.
* ECOG performance status of 0 or 1.
* Participants recruited specifically for PD evaluation must have at least 1 tumour suitable for paired biopsies and be willing to consent to pre-treatment and on-treatment biopsies.

Exclusion Criteria:

* Major surgery within 4 weeks of the first dose of study intervention.
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study intervention.
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study intervention.
* Any known history of persisting severe pancytopenia due to any cause.
* Spinal cord compression unless asymptomatic, treated and stable and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent for at least 4 weeks prior to start of study intervention.
* History of uncontrolled seizures or with need for concurrent administration of more than 2 antiepileptic drugs, or history of epileptic disorder or any seizure history unrelated to tumour.
* History of severe brain injury or stroke.
* Any evidence of severe or uncontrolled systemic diseases including active bleeding diatheses, active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
* Uncontrolled intercurrent illness within the last 12 months.
* Any known predisposition to bleeding.
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD9574.
* Known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s).
* Known contra-indication to gadolinium-enhanced Magnetic Resonance Imaging (MRI) or, if applicable, not able to be maintained on a stable or decreasing dose of corticosteroid regimen (no increase for 7 days) prior to the baseline MRI.
* Any concurrent anti-cancer therapy or concurrent use of prohibited medications.

Module 1:

Part A:

* Have received > one prior line of therapy in any setting with a PARPi-based regimen.
* Participants with an INR >1.5 unless the patient is receiving non-vitamin K antagonist oral anticoagulants.
* Participants with leptomeningeal disease (LMD) unless the LMD is of low volume or is previously treated and the participant is asymptomatic or minimal symptoms.
* Participants with insulin-dependent diabetes.
* Currently on ARA treatment.

Part B:

* Participants with an International Normalised Ratio (INR) >1.5 unless the patient is receiving non-vitamin K antagonist oral anticoagulants.
* Participants with LMD are excluded unless the LMD is of low volume or is previously irradiated and the participant is asymptomatic from the LMD.

Module 2:

* Received a PARPi previously.
* Known hypersensitivity to TMZ or dacarbazine or known history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD9574.
* Have received > 1 prior line of alkylating chemotherapy regimen. Participants who have received procarbazine, lomustine (CCNU), vincristine (PCV) as a prior line of treatment are not allowed.
* Previously experienced Grade 4 haematological toxicities or Grade 3 neutropenia associated with infections, or Grade 3 thrombocytopenia with clinically significant bleeding during prior alkylating chemotherapy.
* Received bevacizumab within the last 6 months.
* Not requiring continuous corticosteroids at a dose of >10 mg prednisone/day or equivalent for at least 4 weeks prior to start of study intervention.

Module 3:

All Panels

* Positive Allen's test
* BMI > 30.0 kg/m2 or body weight > 100.0 kg
* Suffer from claustrophobia.
* Implanted metal devices or implants containing metal.
* An INR >1.5
* Taking acid-reducing agents.

Panel 1

* Received > 1 prior line of therapy in any setting with a PARPi-based regimen
* Participants with LMD

Panel 2

* Received a PARPi previously.
* Known hypersensitivity to TMZ.
* Received > 1 prior line of alkylating chemotherapy regimen.
* Previously experienced Grade 4 haematological toxicities or Grade 3 neutropenia associated with infections, or Grade 3 thrombocytopenia with clinically significant bleeding during prior alkylating chemotherapy.
* Received bevacizumab within the last 6 months.

Panel 3

* Received > one prior line of therapy in any setting with a PARPi-based regimen.
* Participants with LMD.

Module 4:

All participants:

* Current or prior use of immunosuppressive medication within 14 days before the first dose of T-DXd and within 4 weeks for continuous corticosteroids at a dose of approximately > 10 mg prednisone/day or equivalent.
* Should not have received more than 2 prior lines of systemic cytotoxic therapy.
* Prior treatment with HER2 directed TOPO1i ADCs and prior AZD9574 is not permitted.
* Must not enter the study if they received chloroquine/hydroxychloroquine < 14 days prior to the first dose.
* Presence of unresolved toxicities from previous anti-cancer therapy, defined as toxicities not yet resolved to Grade ≤ 1 or baseline.
* Known history of prior platelet transfusion(s) or febrile neutropenia in the advanced disease treatment setting.
* Medical history of myocardial infarction. Participants with troponin levels above ULN at screening and without any myocardial related symptoms.
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or suspected ILD/pneumonitis.
* Additional lung-related exclusion criteria: (a) Lung-specific intercurrent clinically significant illnesses (b) Any autoimmune, connective tissue or inflammatory disorders (c) Prior pneumonectomy.
* Pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy.
* Known hypersensitivity to T-DXd, any of the excipients or other mAbs.
* History of another primary malignancy.
* An uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
* Active primary immunodeficiency, known uncontrolled active HIV infection or active hepatitis B or hepatitis C infection.

Part A (dose escalation):

- Participants with brain metastases are excluded unless asymptomatic, treated, and participant is clinically stable and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent for at least 4 weeks prior to study intervention.

Part B (dose expansion):

- Prior systemic cytotoxic-containing treatment in the metastatic/locally advanced unresectable setting.

Part B (dose expansion) - Participants with Brain Metastases:

* Known and symptomatic leptomeningeal disease.
* Spinal cord compression.

Module 5:

* Current or prior use of immunosuppressive medication within 14 days before the first dose of Dato-DXd and within 4 weeks for continuous corticosteroids at a dose of approximately > 10 mg prednisone/day or equivalent.
* Corticosteroid mouthwash formulations are permitted to prevent and manage certain AEs.
* Prior anti-cancer treatments:

  1. Should not have received more than 2 prior lines of systemic cytotoxic therapy
  2. Prior treatment with PARPi is permitted
  3. Prior TOPO1 inhibitor therapy is NOT permitted
  4. Prior treatment with TROP2-directed ADCs is NOT permitted.
  5. Prior radiation therapy requires the washout periods.
* Must not enter the study if they received chloroquine / hydroxychloroquine < 14 days prior to the first dose.
* History of another primary malignancy.
* History of non-infectious ILD/pneumonitis including radiation pneumonitis that required steroids, has current or suspected ILD/pneumonitis.
* Clinically severe pulmonary function compromise.
* Clinically significant corneal disease.
* History of severe hypersensitivity reactions to Dato-DXd, any of the excipients or to other mabs.
* Participant is pregnant or breastfeeding or planning to become pregnant.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2027-08-11 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs), and Serious Adverse Events (SAEs) | From first dose to post-treatment follow-up (approximately three years)
  The safety and tolerability of AZD9574 as monotherapy and in combination with anti-cancer agents and TMZ in participants with advanced malignancies will be assessed.
Changes from baseline in laboratory findings, electrocardiograms (ECGs), and vital signs | From last assessment prior to first dose to post-treatment follow up visit (approximately three years)
  The safety and tolerability of AZD9574 as monotherapy and in combination with anti-cancer agents and TMZ in participants with advanced malignancies will be assessed.
Change from baseline Eastern Cooperative Oncology Group performance status (ECOG PS) | From last assessment prior to first dose to post-treatment follow up visit (approximately three years)
  The performance status of ECOG will be assessed based on an ECOG grade of 0 to 4 where '0' is a high grade while '4' is a low grade. An ECOG grade of '0' means that the participant is fully active, able to carry on all pre-disease performance without restriction. An ECOG grade of '4' means that the participant is completely disabled, cannot carry on any self-care, and is totally confined to a bed or chair.
Incidence of Dose Limiting Toxicities (DLTs) | Cycle 0 and Cycle 1 (Day 1 to Day 35)
  The safety and tolerability of AZD9574 as monotherapy and in combination with anti-cancer agents in participants with advanced malignancies will be assessed at each dose level.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) | Cycle 0, Cycle 1 Day 1, Cycle 1 Day 16 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The AUC of AZD9574 following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents will be evaluated.
Maximum plasma concentration (Cmax) | Cycle 0, Cycle 1 Day 1, Cycle 1 Day 16 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The Cmax of AZD9574 following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents will be evaluated.
Time to reach maximum plasma concentration (tmax) | Cycle 0, Cycle 1 Day 1, Cycle 1 Day 16 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The tmax of AZD9574 following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents will be evaluated.
Minimum plasma concentration at steady state (Cmin,ss) | Cycle 0, Cycle 1 Day 1, Cycle 1 Day 16 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The Cmin,ss of AZD9574 following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents will be evaluated.
Half-life (t1/2) | Cycle 0, Cycle 1 Day 1, Cycle 1 Day 16 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The t1/2 of AZD9574 following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents will be evaluated.
Accumulation ratio | Cycle 0, Cycle 1 Day 1, Cycle 1 Day 16 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The accumulation ratio of AZD9574 following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents will be evaluated.
Dose proportionality | Cycle 0, Cycle 1 Day 1, Cycle 1 Day 16 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The dose proportionality of AZD9574 following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents will be evaluated.
Module 1: Assessment of pH2AX (phospho-histone 2AX) (Ser139) PD biomarker modulations | Screening, Cycle 0 Day 1, Cycle 1 Day 8, and Cycle 1 day 15 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The PD biomarker modulations of pH2AX (Ser139) at baseline and during treatment or pre-treatment will be assessed in tumour tissue when given orally as monotherapy.
Module 1: Percentage change in target lesion (TL) size | From Baseline to every 8 weeks until disease progression (approximately three years)
  The percentage change in TL size will be determined for participants with measurable disease at baseline and is derived at each visit.
Module 1: Objective Response Rate (ORR) | From Baseline to every 8 weeks until disease progression (approximately three years)
  ORR is defined as the percentage of participants who have a confirmed response of Complete Response (CR) or Partial Response (PR) prior to any evidence of progression according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1) for solid tumours, RECIST v1.1 and/or Prostate Cancer Working Group 3 (PCWG3 [bone]) for prostate cancer, and Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) for brain metastases.
Module 1: Duration of Response (DoR) | First documented response until the date of documented progression or end of study (approximately three years)
  The DoR is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of disease progression according to RECIST v1.1 for solid tumours, RECIST v1.1 and/or PCWG3 for prostate cancer, and RANO-BM for brain metastases.
Module 1: Time To Response (TTR) | From the first dose until the first documentation of a subsequently confirmed objective response (approximately three years)
  TTR is defined as the time from first dose until the first documentation of a subsequently confirmed objective response according to RECIST v1.1 for solid tumours, RECIST v1.1 and/or PCWG3 for prostate cancer, and RANO-BM for brain metastases.
Module 1: Progression Free Survival (PFS)/radiographic Progression-Free Survival (rPFS) | From the start of first treatment until the date of objective disease progression or death (approximately three years)
  PFS and rPFS are defined as the time from start of first treatment until the date of objective disease progression or death regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy prior to progression according to RECIST v1.1 for solid tumours, RECIST v1.1 and/or PCWG3 for prostate cancer, and RANO-BM for brain metastases.
Module 1: Cancer Antigen 125 (CA125) response evaluated according to the GCIG criteria (for ovarian patients only) | From Screening until disease progression or death (approximately three years)
  CA125 response is defined as at least a 50% reduction in CA125 levels from a pre-treatment sample.
Module 1: Proportion of participants achieving a ≥ 50% decrease in PSA from baseline to the lowest post-baseline PSA result (for prostate cancer only) | From screening until disease progression or death (approximately three years)
  PSA50 response is defined as the proportion of participants achieving a ≥ 50% decrease in Prostate Specific Antigen (PSA) from baseline to the lowest post-baseline PSA, confirmed by a consecutive PSA at least 3 weeks later and will be based on PSA evaluable participants.
Module 1: Radiological response evaluated according to RECIST v1.1 + Prostate Cancer Working Group 3 (PCWG3) response evaluation criteria (for prostate cancer only) | Up to the End Of Trial (EOT) [approximately three years]
  In participants with prostate cancer, disease progression will be deemed to have occurred if soft tissue disease progression, bone lesion progression, or death are met.
Module 1 (Food effect): AUC | Cycle 0 Day 1,2,3, Cycle 1 Day 1,2,8 to 15 and Cycle 2 Day 1, and Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To investigate the effect of a high-fat meal on the AUC of AZD9574 (Fasted and fed state).
Module 1 (Food effect) : Area under the curve from 0 to t [AUC (0-t)] | Cycle 0 Day 1,2,3, Cycle 1 Day 1,2,8 to 15 and Cycle 2 Day 1, and Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To investigate the effect of a high-fat meal on the AUC (0-t) of AZD9574 (Fasted and fed state).
Module 1 (Food effect): Cmax | Cycle 0 Day 1,2,3, Cycle 1 Day 1,2,8 to 15 and Cycle 2 Day 1, and Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To investigate the effect of a high-fat meal on the Cmax of AZD9574 (Fasted and fed state).
Module 1 (Food effect): Tmax | Cycle 0 Day 1,2,3, Cycle 1 Day 1,2,8 to 15 and Cycle 2 Day 1, and Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To investigate the effect of a high-fat meal on the Tmax of AZD9574 (Fasted and fed state).
Module 1 (Food effect) : Maximum plasma concentration (Cmax) ratio (with /without a high fat meal) | Cycle 0 Day 1,2,3, Cycle 1 Day 1,2,8 to 15 and Cycle 2 Day 1, and Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To investigate the effect of a high-fat meal on the Cmax ratio of AZD9574 (Fasted and fed state).
Module 1 (ARA effect): AUC | Cycle 0 Day 1,3, Cycle 1 Day 1,2,8 to 15,16, Cycle 2 Day 1, Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To assess the effect of famotidine on the AUC of AZD9574 (with and without famotidine).
Module 1 (ARA effect): AUC (0-t) | Cycle 0 Day 1,3, Cycle 1 Day 1,2,8 to 15,16, Cycle 2 Day 1, Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To assess the effect of famotidine on the AUC (0-t) of AZD9574 (with and without famotidine).
Module 1 (ARA effect): Cmax | Cycle 0 Day 1,3, Cycle 1 Day 1,2,8 to 15,16, Cycle 2 Day 1, Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To assess the effect of famotidine on the Cmax of AZD9574 (with and without famotidine).
Module 1 (ARA effect): Tmax | Cycle 0 Day 1,3, Cycle 1 Day 1,2,8 to 15,16, Cycle 2 Day 1, Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To assess the effect of famotidine on the Tmax of AZD9574 (with and without famotidine).
Module 1 (ARA effect) : Cmax ratio (with /without famotidine) | Cycle 0 Day 1,3, Cycle 1 Day 1,2,8 to 15,16, Cycle 2 Day 1, Cycle 3 Day 1 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  To assess the effect of famotidine on the Cmax ratio of AZD9574 (with and without famotidine).
Module 2: Percentage change in TL size | From Baseline to every 8 weeks until objective disease progression (approximately three years)
  The percentage change in TL size will be determined for participants with measurable disease at baseline and is derived at each visit by the measurability of TL according to Response Assessment in Neuro-Oncology - high-grade glioma (RANO-HGG) or Response Assessment in Neuro-Oncology - low-grade glioma (RANO-LGG).
Module 2: ORR | From Baseline to every 8 weeks until objective disease progression (approximately three years)
  The ORR is defined as the percentage of participant with high- or low-grade gliomas with at least one visit response of CR or PR according to RANO-HGG or RANO-LGG.
Module 2: DoR | First documented response until the date of documented progression or end of study (approximately three years)
  The DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression according to RANO-HGG or RANO-LGG.
Module 2: TTR | First dose until the first documentation of a subsequently confirmed objective response (approximately three years)
  TTR is defined as the time from first dose until the first documentation of a subsequently confirmed objective response according to RANO-HGG or RANO-LGG.
Module 2: PFS | From the start of first treatment until the date of objective disease progression or death (approximately three years)
  The PFS is defined as the time from the start of study intervention until the date of objective disease progression or death regardless of whether the participant withdraws from study intervention or receives another anti-cancer therapy prior to progression according to RANO-HGG or RANO-LGG.
Module 3: Occupancy | From Screening to Cycle 2 Day 1
  Occupancy (%) is defined as the estimated difference in radioligand binding to PARP1 from baseline to PET examination after drug administration.
Module 3: Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose to post-treatment follow-up (approximately three years)
  The safety of radioligand [11C]AZ14193391 will be assessed.
Module 3: AUC | Cycle 0 Day 1 & 5, Cycle 1 Day 5 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The AUC of AZD9574 following single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with TMZ will be evaluated.
Module 3: Cmax | Cycle 0 Day 1 & 5, Cycle 1 Day 5 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The Cmax of AZD9574 following single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with TMZ will be evaluated.
Module 3: tmax | Cycle 0 Day 1 & 5, Cycle 1 Day 5 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The tmax of AZD9574 following single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with TMZ will be evaluated.
Module 3: Cmin,ss | Cycle 0 Day 1 & 5, Cycle 1 Day 5 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The Cmin,ss of AZD9574 following single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with TMZ will be evaluated.
Module 3: t1/2 | Cycle 0 Day 1 & 5, Cycle 1 Day 5 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The t1/2 of AZD9574 following single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with TMZ will be evaluated.
Module 3: Accumulation ratio | Cycle 0 Day 1 & 5, Cycle 1 Day 5 (Cycle 0 = 7 days; Cycle 1 = 28 days)
  The accumulation ratio of AZD9574 following single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with TMZ will be evaluated.
Module 3: Percentage change in target lesion (TL) size | From Baseline to every 8 weeks until disease progression (approximately three years)
  The percentage change in TL size will be determined for participants with measurable disease at baseline and is derived at each visit.
Module 3: ORR | From Baseline to every 8 weeks until disease progression (approximately three years)
  ORR is defined as the percentage of participants who have a confirmed response of Complete Response (CR) or Partial Response (PR) prior to any evidence of progression according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1) for solid tumours, RECIST v1.1 and/or Prostate Cancer Working Group 3 (PCWG3 [bone]) for prostate cancer, and Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) for brain metastases and according to Response Assessment in Neuro-Oncology - high-grade glioma (RANO-HGG) or Response Assessment in Neuro-Oncology - low-grade glioma (RANO-LGG).
Module 3: DoR | First documented response until the date of documented progression or end of study (approximately three years)
  The DoR is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of disease progression according to RECIST v1.1 for solid tumours, RECIST v1.1 and/or PCWG3 for prostate cancer, RANO-BM for brain metastases and RANO-HGG or RANO-LGG.
Module 3: TTR | From the first dose until the first documentation of a subsequently confirmed objective response (approximately three years)
  TTR is defined as the time from first dose until the first documentation of a subsequently confirmed objective response according to RECIST v1.1 for solid tumours, RECIST v1.1 and/or PCWG3 for prostate cancer, RANO-BM for brain metastases and RANO-HGG or RANO-LGG.
Module 3: Cancer Antigen 125 (CA125) response evaluated according to the GCIG criteria (for ovarian patients only) | From Screening until disease progression or death (approximately three years)
  CA125 response is defined as at least a 50% reduction in CA125 levels from a pre-treatment sample.
Module 3: Proportion of participants achieving a ≥ 50% decrease in PSA from baseline to the lowest post-baseline PSA result (for prostate cancer only) | From screening until disease progression or death (approximately three years)
  PSA50 response is defined as the proportion of participants achieving a ≥ 50% decrease in Prostate Specific Antigen (PSA) from baseline to the lowest post-baseline PSA, confirmed by a consecutive PSA at least 3 weeks later and will be based on PSA evaluable participants.
Module 3: Progression Free Survival (PFS)/radiographic Progression-Free Survival (rPFS) | From the start of first treatment until the date of objective disease progression or death (approximately three years)
  PFS and rPFS are defined as the time from start of first treatment until the date of objective disease progression or death regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy prior to progression according to RECIST v1.1 for solid tumours, RECIST v1.1 and/or PCWG3 for prostate cancer, RANO-BM for brain metastases and RANO-HGG or RANO-LGG.
Module 3: Radiological response evaluated according to RECIST v1.1 + Prostate Cancer Working Group 3 (PCWG3) response evaluation criteria (for prostate cancer only) | Up to the End Of Trial (EOT) [approximately three years]
  In participants with prostate cancer, disease progression will be deemed to have occurred if soft tissue disease progression, bone lesion progression, or death are met.
Module 4 : AUC | AZD9574 (Parts A and B): Cycle (C) 1 Day (D) X1 (first dose), X2 (last dose), C2 D1, X1 (first dose), D15 (part A only), and C3 D1 T DXd: C1 D1, X1 (pre-dose AZD9574), X2, C2 D1, C3 D1, and C4 D1, up to safety follow-up (40-days after last dose)
  To characterise the AUC of AZD9574, T-DXd following a single dose and at steady state after multiple dosing, when given in combination with T-DXd.
Module 4 : Cmax | AZD9574 (Parts A and B): C1 X1 (first dose), X2 (last dose), C2 D1, X1 (first dose), D15 (part A only), and C3 D1 T DXd: C1 D1, X1 (pre-dose AZD9574), X2, C2 D1, C3 D1, and C4 D1, up to safety follow-up (40-days after last dose)
  To characterise the Cmax of AZD9574, T-DXd following a single dose and at steady state after multiple dosing, when given in combination with T-DXd.
Module 4 : Tmax | AZD9574 (Parts A and B): C1 X1 (first dose), X2 (last dose), C2 D1, X1 (first dose), D15 (part A only), and C3 D1 T DXd: C1 D1, X1 (pre-dose AZD9574), X2, C2 D1, C3 D1, and C4 D1, up to safety follow-up (40-days after last dose)
  To characterise the Tmax of AZD9574, T-DXd following a single dose and at steady state after multiple dosing, when given in combination with T-DXd.
Module 4 : Assessment of pH2AX (phospho-histone 2AX) (Ser139) PD biomarker modulations | Cycle 1 Day X1, Day X2 [last of AZD9574 dosing] (Cycle 1 = 28 days)
  To characterise the PD of AZD9574 in tumour tissue, following a single dose and at steady state after multiple dosing, when given orally in combination with T-DXd.
Module 4 : Presence of ADAs for T-DXd | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Safety follow-up (FU) 40 [+ 7] days after last dose
  To investigate the immunogenicity of T-DXd.
Module 4 : Incidence of Adverse event of special interest (AESI) | From first dose until the safety FU (40 [+ 7] days) after discontinuation
  To monitor risks associated with T-DXd (AESI) in study participants.
Module 4 (Part A): ORR | From Baseline to every 6 weeks until disease progression (approximately three years)
  ORR is defined as the percentage of participants who have a confirmed response of Complete Response (CR) or Partial Response (PR) prior to any evidence of progression according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1).
Module 4 (Part B): ORR | From Baseline to every 6 weeks for the first 24 weeks and then every 9 weeks until disease progression (approximately three years)
  ORR is defined as the percentage of participants who have a confirmed response of CR or PR prior to any evidence of progression according to RECIST v1.1, RECIST v1.1 and RANO-BM for participants with brain metastasis.
Module 4 (Part A): DoR | First documented response until the date of documented progression or end of study (approximately three years)
  The DoR is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of disease progression according to RECIST v1.1.
Module 4 (Part B): DoR | First documented response until the date of documented progression or end of study (approximately three years)
  The DoR is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of disease progression according to RECIST v1.1, RECIST v1.1 and RANO-BM for participants with brain metastasis.
Module 4 (Part A): PFS | From the start of first treatment until the date of objective disease progression or death (approximately three years)
  PFS is defined as the time from start of first treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy prior to progression according to RECIST v1.1.
Module 4 (Part B): PFS | From the start of first treatment until the date of objective disease progression or death (approximately three years)
  PFS is defined as the time from start of first treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy prior to progression according to RECIST v1.1, RECIST v1.1 and RANO-BM for participants with brain metastasis.
Module 4 (Part A): TTR | From the first dose until the first documentation of a subsequently confirmed objective response (approximately three years)
  TTR is defined as the time from first dose until the first documentation of a subsequently confirmed objective response according to RECIST v1.1.
Module 4 (Part B): TTR | From the first dose until the first documentation of a subsequently confirmed objective response (approximately three years)
  TTR is defined as the time from first dose until the first documentation of a subsequently confirmed objective response according to RECIST v1.1, RECIST v1.1 and RANO-BM for participants with brain metastasis.
Module 4 (Part B only): Progression-free survival at 6 months (PFS6) | At 6 months after start of first treatment
  The PFS is defined as the time from the start of study intervention until the date of objective disease progression or death regardless of whether the participant withdraws from study intervention or receives another anti-cancer therapy prior to progression according to RECIST v1.1, RECIST v1.1 and RANO-BM for participants with brain metastasis.
Module 4 (Part B): Number of participants experiencing each level of symptomatic AEs as measured by the Patient-Reported Outcomes Version of the common terminology criteria for adverse events (PRO-CTCAE) (participants without brain metastases only) | From the first dose until the end of 12 months or EOT, whichever comes first (approximately three years)
  The PRO-CTCAE is an item library of symptoms experienced by participants while undergoing treatment of their cancer. It assess the presence/absence, severity, frequency, and interference of treatment-related symptoms from the participant's perspective.
Module 4 (Part B): Number of participants reporting overall side effect bother on the patient's global impression of treatment tolerability (PGI-TT) while receiving treatment (participants without brain metastases only) | From the first dose until the end of 12 months or EOT, whichever comes first (approximately three years)
  The PGI-TT is a single item assessment of the participant's overall level of bother due to treatment-related side effects of cancer treatment over a 1-week period.
  Participants will be asked to choose the response that best describes the severity of their overall cancer symptoms over the past week to aid in the interpretation of other clinical outcomes and explore the cumulative impact of treatment-related side effects. The response options are: "not at all", "a little bit", "somewhat", "quite a bit", and "very much".
Module 4: Cancer Antigen 125 (CA125) response evaluated according to the GCIG criteria (for ovarian patients only) | From Screening until disease progression or death (approximately three years)
  CA125 response is defined as at least a 50% reduction in CA125 levels from a pre-treatment sample.
Module 5 : AUC | AZD9574: Cycle 1 Day X1 (first dose), X2 (last dose), Cycle 2 Day 1, X1 (first dose), Day 15, Cycle 3 Day 1 Dato-DXd: Cycle 1 Day 1, X1 (pre-dose AZD9574), X2, Cycle 2 Day 1, Cycle 4 Day 1, C8D1, every 4 cycles thereafter on Day 1
  To assess the AUC of AZD9574 and Dato-DXd.
Module 5 : Cmax | AZD9574: Cycle 1 Day X1 (first dose), X2 (last dose), Cycle 2 Day 1, X1 (first dose), Day 15, Cycle 3 Day 1 Dato-DXd: Cycle 1 Day 1, X1 (pre-dose AZD9574), X2, Cycle 2 Day 1, Cycle 4 Day 1, C8D1, every 4 cycles thereafter on Day 1
  To assess the Cmax of AZD9574 and Dato-DXd.
Module 5 : Tmax | AZD9574: Cycle 1 Day X1 (first dose), X2 (last dose), Cycle 2 Day 1, X1 (first dose), Day 15, Cycle 3 Day 1 Dato-DXd: Cycle 1 Day 1, X1 (pre-dose AZD9574), X2, Cycle 2 Day 1, Cycle 4 Day 1, C8D1, every 4 cycles thereafter on Day 1
  To assess the Tmax of AZD9574 and Dato-DXd.
Module 5 : Assessment of pH2AX (phospho-histone 2AX) (Ser139) PD biomarker modulations | Cycle 1 Day X1, Day X2 [last of AZD9574 dosing] (Cycle 1 = 28 days)
  To characterise the PD of AZD9574 in tumour tissue, following a single dose and at steady state after multiple dosing, when given orally in combination with Dato-DXd.
Module 5 : Presence of positive ADAs for Dato-DXd | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, EoT(End of treatment) ± 7 days, Safety follow up (FU) 28 [+ 7] days after last dose
  To investigate the immunogenicity of Dato-DXd.
Module 5: ORR | From Baseline to every 6 weeks until disease progression (approximately three years)
  ORR is defined as the percentage of participants who have a confirmed response of Complete Response (CR) or Partial Response (PR) prior to any evidence of progression according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1) and PCWG3 for prostate cancer.
Module 5: DoR | First documented response until the date of documented progression or end of study (approximately three years)
  The DoR is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of disease progression according to RECIST v1.1.
Module 5: TTR | From the first dose until the first documentation of a subsequently confirmed objective response (approximately three years)
  TTR is defined as the time from first dose until the first documentation of a subsequently confirmed objective response according to RECIST v1.1.
Module 5: Progression Free Survival (PFS)/radiographic Progression-Free Survival (rPFS) | From the start of first treatment until the date of objective disease progression or death (approximately three years)
  PFS and rPFS are defined as the time from start of first treatment until the date of objective disease progression or death regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy prior to progression according to RECIST v1.1 for solid tumours, RECIST v1.1 and/or PCWG3 for prostate cancer.
Module 5 : Incidence of AESIs | From first dose until the safety FU (40 [+ 7] days) after discontinuation
  To describe the prevalence (or incidence/frequency, etc) of Dato-DXd AESIs in study participants.
Module 5: Cancer Antigen 125 (CA125) response evaluated according to the GCIG criteria (for ovarian patients only) | From Screening until disease progression or death (approximately three years)
  CA125 response is defined as at least a 50% reduction in CA125 levels from a pre-treatment sample.
Module 5: Proportion of participants achieving a ≥ 50% decrease in PSA from baseline to the post-baseline PSA result (for prostate cancer only) | From screening until disease progression or death (approximately three years)
  PSA50 response is defined as the proportion of participants achieving a ≥ 50% decrease in Prostate Specific Antigen (PSA) from baseline to the lowest post-baseline PSA, confirmed by a consecutive PSA at least 3 weeks later and will be based on PSA evaluable participants.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (10):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
- Australia (4):
  - Research Site, Camperdown
  - Research Site, Darlinghurst
  - Research Site, Melbourne
  - Research Site, Randwick
- Germany (4):
  - Research Site, Bayern
  - Research Site, Berlin
  - Research Site, Heidelberg
  - Research Site, Mainz
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Málaga
  - Research Site, Pozuelo de Alarcón
  - Research Site, Sant Cugat del Vallès
  - Research Site, Seville
- Sweden (2):
  - Research Site, Lund
  - Research Site, Stockholm
- United Kingdom (3):
  - Research Site, Glasgow, Scotland
  - Research Site, London
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Staniszewska AD, Pilger D, Gill SJ, Jamal K, Bohin N, Guzzetti S, Gordon J, Hamm G, Mundin G, Illuzzi G, Pike A, McWilliams L, Maglennon G, Rose J, Hawthorne G, Cortes Gonzalez M, Halldin C, Johnstrom P, Schou M, Critchlow SE, Fawell S, Johannes JW, Leo E, Davies BR, Cosulich S, Sarkaria JN, O'Connor MJ, Hamerlik P. Preclinical Characterization of AZD9574, a Blood-Brain Barrier Penetrant Inhibitor of PARP1. Clin Cancer Res. 2024 Apr 1;30(7):1338-1351. doi: 10.1158/1078-0432.CCR-23-2094. PMID 37967136
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/347358